CLINICAL TRIAL: NCT04543422
Title: Green Tea Extracts for Mild-to-moderate Diabetic Peripheral Neuropathy A Randomized Controlled Trial
Brief Title: Green Tea Extracts for Mild-to-moderate Diabetic Peripheral Neuropathy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Egyptian Biomedical Research Network (Network)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: EBRN298
Record Dates: First submitted 2020-08-29; First posted 2020-09-10 (Actual); Last update posted 2020-09-10 (Actual); Status verified 2020-08

CONDITIONS: Diabetic Peripheral Neuropathy
MeSH Terms: interventions — Tea

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Green tea extracts (Experimental): Patients in this arm received green tea extract capsules
  Interventions: Dietary Supplement: Green tea
- Placebo (Placebo Comparator): Patients in this arm received placebo treatment
  Interventions: Other: Placebo

INTERVENTIONS:
Dietary Supplement: Green tea — Green tea extract capsules
  Arms: Green tea extracts
Other: Placebo — Placebo containing inert material.
  Arms: Placebo

SUMMARY:
the present randomized placebo-controlled study aimed to evaluate the effect of green tea extract administration on the clinical and neurophysiological parameters in patients with mild-to-moderate diabetic peripheral neuropathy.

ELIGIBILITY:
Inclusion Criteria:

* Diabetic patients with peripheral neuropathy

Exclusion Criteria:

* Patients under treatment of diabetic peripheral neuropathy.
* Patients with other causes of peripheral neuropathy.

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Actual)
Dates: Start 2019-01-01 (Actual); Primary Completion 2020-03-01 (Actual); Study Completion 2020-03-01 (Actual)

PRIMARY OUTCOMES:
Toronto Clinical Scoring System | three months
  Improvement describes the difference between baseline and post-intervention outcome parameters

CONTACTS AND LOCATIONS:
Locations (1):
- Al-Azhar University Faculty of Medicine, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No